CLINICAL TRIAL: NCT00005077
Title: Phase I Study of Oxaliplatin in Patients With Advanced Malignancies and Varying Degrees of Liver Dysfunction (Summary Last Modified 04/2000)
Brief Title: Oxaliplatin in Treating Patients With Advanced Cancer Plus Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067684; U01CA062505 (NIH); R03CA080647 (NIH); P30CA033572 (NIH); CHNMC-PHI-26; CHNMC-IRB-99108; NCI-00-C-0172; NCI-NMOB-B00-033; PCI-99105; NCI-T99-0050
Record Dates: First submitted 2000-04-06; First posted 2004-04-12 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of oxaliplatin in treating patients who have advanced cancer plus liver dysfunction.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of oxaliplatin in patients with advanced malignancies and varying degrees of liver dysfunction. II. Determine the effects of hepatic dysfunction on the plasma pharmacokinetics and pharmacodynamics of oxaliplatin in these patients.

OUTLINE: This is a dose escalation, multicenter study. Patients are stratified according to liver function as defined by the following: Group A: Normal liver function - Bilirubin, SGOT, and alkaline phosphatase no greater than upper limit of normal (ULN) Group B: Mild liver dysfunction - Bilirubin no greater than ULN; SGOT greater than ULN to 2.5 times ULN and/or alkaline phosphatase greater than ULN to 5 times ULN Group C: Moderate liver function - Bilirubin greater than ULN to 3.0 mg/dL and/or SGOT greater than 2.5 times ULN and/or alkaline phosphatase greater than 5 times normal Group D: Severe liver dysfunction - Bilirubin greater than 3.1 mg/dL and any SGOT or alkaline phosphatase Group E: Patients who have received a liver transplant Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients in groups B, C, and D receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose- limiting toxicity.

PROJECTED ACCRUAL: Approximately 72 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or unresectable malignancy for which no curative or palliative treatment exists No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 2 months Hematopoietic: Platelet count at least 100,000/mm3 WBC at least 3,000/mm3 OR Absolute neutrophil count at least 1,500/mm3 Hepatic: Abnormal liver function allowed Renal: Creatinine normal OR Creatinine clearance at least 60 mL/min Cardiovascular: No symptomatic congestive heart failure No unstable angina pectoris No cardiac arrhythmia Other: No clinically significant neuropathy Not pregnant or nursing Fertile patients must use effective contraception No history of allergy to platinum compounds or antiemetics which may be used with study No uncontrolled concurrent illness (e.g., ongoing or active infection)

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent colony stimulating factors during first course of study Chemotherapy: No more than 3 prior regimens of chemotherapy At least 6 weeks since prior platinum chemotherapy At least 4 weeks since other prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to more than 30% of bone marrow Surgery: At least 10 days since placement of biliary shunt Other: No other concurrent investigational agents No concurrent antiretroviral therapy (HAART) in HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02

CONTACTS AND LOCATIONS:
Overall Officials: James H. Doroshow, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (11):
- United States (11):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin